CLINICAL TRIAL: NCT00941694
Title: Asthma Self-Management in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Alan Baptist, Assistant Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: N011060
Record Dates: First submitted 2009-07-17; First posted 2009-07-20 (Estimated); Last update posted 2013-01-16 (Estimated); Status verified 2013-01

CONDITIONS: Asthma; Aged
Keywords: asthma; aged; self care
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Self-Management Intervention (Experimental): Will receive 6 asthma self-management group or individual session over a 7 week period
  Interventions: Behavioral: Self management intervention
- Control (Placebo Comparator): Group will receive 3 phone calls not related to asthma self management over a 7 week period
  Interventions: Behavioral: placebo group

INTERVENTIONS:
Behavioral: Self management intervention — Intervention arm will receive 6 group or individual sessions over a 7 week period
  Arms: Self-Management Intervention
Behavioral: placebo group — 3 phone calls not related to asthma self-management
  Arms: Control

SUMMARY:
Asthma self-management is an effective way to improve the outcomes of patients with asthma. However, to be most effective these interventions should be targeted and designed toward a specific population or group. There is currently no asthma self-management intervention directed towards older adults. The hypothesis is that a 6-session asthma self-management intervention will improve the outcomes of older patients with asthma.

ELIGIBILITY:
Inclusion Criteria:: Age over 65, physician diagnosed asthma, need for daily asthma control medication, access to a telephone.

-

Exclusion Criteria: Smoking history greater than 40 pack years, current smoker, mental impairment that would preclude participation in the asthma self management program

-

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 70 (Actual)
Dates: Start 2009-07; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Asthma Quality of Life Questionnaire | 3 months, 6 months, 1 year

SECONDARY OUTCOMES:
Asthma Control Questionnaire | 3 months, 6 months, 12 months
Health Care Utilization | 3 months, 6 months, 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Alan P Baptist, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States